CLINICAL TRIAL: NCT01535287
Title: The Effect of Intramuscular Dexmedetomidine on Emergence Agitation in Children Undergoing With or Without Tube Insertion Under General Anesthesia
Brief Title: Effect of Dexmedetomidine on Emergence Agitation in Children With or Without Tube Insertion Under General Anesthesia
Status: Completed | Phase: Phase 4 | Type: Interventional
Sponsor: Martin Mueller (Other)
Responsible Party: Sponsor-Investigator, Martin Mueller, Principal Investigator, University of Iowa
Organization: University of Iowa (Other)
Allocation: Randomized | Model: Parallel | Masking: Triple | Purpose: Treatment
Other Study IDs: 201006723
Record Dates: First submitted 2012-01-20; First posted 2012-02-17 (Estimated); Results first posted 2018-07-09 (Actual); Last update posted 2018-07-09 (Actual); Status verified 2018-06

CONDITIONS: Myringotomy
Keywords: Dexmedetomidine; Emergence Agitation; Myringotomy; Children; General Anesthesia
MeSH Terms: conditions — Emergence Delirium | interventions — Dexmedetomidine

STUDY DESIGN:
Who Masked: Participant, Care Provider, Investigator
Oversight: Data Monitoring Committee: Yes

ARMS (2):
- Dexmedetomidine (Active Comparator): Single injection of Dexmedetomidine (study medication) compared to receiving Placebo in Myringotomy surgery decreases emergence agitation.
  Interventions: Drug: Dexmedetomidine
- Placebo (Placebo Comparator): Single injection of Dexmedetomidine (study medication) compared to receiving Placebo in Myringotomy surgery decreases emergence agitation.
  Interventions: Drug: Dexmedetomidine

INTERVENTIONS:
Drug: Dexmedetomidine — Active study agent: Dexmedetomidine at 1 microgram/kilogram Intramuscular (IM) Placebo study agent: Same volume as the study drug of placebo (normal saline).
  All blinding, labeling, preparation, storage of agents done by the pharmacist. The drug will be administered into the deltoid muscle by using a TB syringe attached to a 3/4 inch length and 25 Gauge width needle by anesthesia provider after the induction of general anesthesia by the anesthesia provider.
  Other Names: Precedex

SUMMARY:
The investigators are inviting your child to participate in this research study because your child is having myringotomy (putting a tiny incision in the eardrum with or without tube insertion) under general anesthesia.

The purpose of this study is to determine whether a single injection of Dexmedetomidine (study medication) decreases the frequency of awaking from anesthesia frightened or agitated in children having myringotomy surgery as compared to those children who receive placebo (sterile saltwater).

DETAILED DESCRIPTION:
Emergence agitation (EA) is common in children, especially in the preschool age group who undergo general anesthesia. It has been described as a mental disturbance during the recovery from general anesthesia and can consist of hallucinations, delusions and confusion in the child. To the parent or caregivers this may be seen as moaning, restlessness, involuntary physical activity & thrashing about in bed. Emergence agitation (EA) can result in the child losing their intravenous therapy (IV) access & bodily injury. Some agitated children may retain vivid memories about their negative experience waking up from anesthesia. This can result in seeing new behaviors by the child such as anxiety, nighttime crying and temper tantrums. Dexmedetomidine given as an injection into the muscle of children is considered investigational, which means it hasn't been approved by the U.S. FDA for treatment of this problem in children.

Immediately following surgery measurements of eye contact, purposeful actions, aware of surroundings, restless and crying are observed and recorded using the Pediatric Anesthesia Emergence Delirium (PAED) scale in PACU.

Follow-up is made approximately 3 days after surgery by phone call or/and email with parent(s) to see if child has experienced any of the following: sleep disturbances, anxiety, eating disturbances, postoperative muscle pain or swelling at the injection site.

ELIGIBILITY:
Inclusion Criteria:

* ASA I or II (American Society of Anesthesiology classification ASA I means patients without systemic disease, ASA II means patients with one controlled systemic medical disease eg: Diabetes, Hypertension.)
* Between the ages of 1 and 10 years
* Undergoing BMT under general anesthesia.

Exclusion Criteria:

* ASA III or higher (Patients with 2 or more medical systemic disease that is not under control, eg: uncontrolled Diabetes)
* Congenital diseases
* Coagulation disorders
* Known allergic reaction to dexmedetomidine
* Serious preexisting impairment of respiratory, cardiovascular, hepatic, renal, neurological or endocrine functions
* Severe upper airway infection
* Predicted difficult airway
* Preexisting psychiatric disorders

Ages: 1 Year to 10 Years | Sex: All | Healthy Volunteers: No
Age Groups: Child
Enrollment: 140 (Actual)
Dates: Start 2011-01-04 (Actual); Primary Completion 2013-10-08 (Actual); Study Completion 2013-10-08 (Actual)

CONTACTS AND LOCATIONS:
Overall Officials: Martin Mueller, M.D., Principal Investigator — University of Iowa Hospital and Clinics
Locations (1):
- University of Iowa Hospital and Clinics, Iowa City, Iowa, United States

IPD SHARING:
Plan to Share IPD: No

RESULTS

PARTICIPANT FLOW:
Groups:
- Dexmedetomidine; Placebo: Single injection of Dexmedetomidine (study medication) compared to receiving Placebo in Myringotomy surgery decreases emergence agitation.
  Dexmedetomidine: Active study agent: Dexmedetomidine at 1 microgram/kilogram Intramuscular (IM) Placebo study agent: Same volume as the study drug of placebo (normal saline).
  All blinding, labeling, preparation, storage of agents done by the pharmacist. The drug will be administered into the deltoid muscle by using a TB syringe attached to a 3/4 inch length and 25 Gauge width needle by anesthesia provider after the induction of general anesthesia by the anesthesia provider.
Period: Overall Study
Arm/Group | Dexmedetomidine | Placebo
Started | 70 | 70
Completed | 65 | 64
Not Completed | 5 | 6
Not completed — drug not prepared in time | 5 | 6

BASELINE CHARACTERISTICS:
Groups:
- Total: Total of all reporting groups
Arm/Group | Dexmedetomidine | Placebo | Total
Number analyzed (Participants) | 65 | 64 | 129
Age, Categorical [Count of Participants; unit: Participants]
  <=18 years | 65 | 64 | 129
  Between 18 and 65 years | 0 | 0 | 0
  >=65 years | 0 | 0 | 0
Age, Continuous [Mean (Standard Deviation); unit: month] | 37 (26) | 39 (30) | 38 (30)
Sex: Female, Male [Count of Participants; unit: Participants]
  Female | 30 | 32 | 62
  Male | 35 | 32 | 67
Region of Enrollment [Number; unit: participants]
  United States | 65 | 64 | 129

OUTCOME MEASURES:

1. Primary Outcome: Participant's Severity of Emergent Agitation (EA) Using the Pediatric Anesthesia Emergence Delirium (PAED) Scale in PACU (Post-Op Area).
Description: The aim/measurement of the study is to determine whether or not a single IM injection of Dexmedetomidine will reduce the severity of Emergent Agitation (EA) in children undergoing Bilateral Myringotomy with/without tubes under general anesthesia.
  We used the only validated scale to assess the severity of post operative emergence delirium in pediatrics. This Pediatric Anesthesia Emergence Delirium (PAED) scale is a composite score of the following items:
  1. Makes eye contact with caregiver.
  2. Child's actions are purposeful.
  3. Child aware of his/her surroundings.
  4. The child is restless.
  5. The child is inconsolable.
  Items 1, 2, and 3 are reversed scored as follows: 4-not at all, 3-a little, 2-quite a bit, 1-very much, 0-extremely. Items 4 and 5 are scored as follows: 0-not at all, 1-a little, 2-quite a bit, 3-very much, 4-extremely.
  The total score will range from 0 to 20; with 0 indicating no emergence delirium and 20 indicating extreme emergence delirium.
Time Frame: Participants will be followed for the duration of first PACU recovery step, an expected average visit of 30 minutes. Measurements will be observed immediately following subject's awakening from anesthesia.
Measure: Mean (Standard Deviation); unit: units on a scale
Arm/Group | Dexmedetomidine | Placebo
Number analyzed (Participants) | 65 | 64
units on a scale | 7 (6) | 8 (6)

2. Secondary Outcome: Duration of Stay in PACU
Description: Duration of stay in the PACU (Post-Op Area) until discharge criteria are met based on modified PADSS score: level of consciousness, physical activity, hemodynamic stability, respiratory stability, oxygen saturation status, post-operative pain, and post-operative emetic symptoms. Duration of time will be measured in total minutes participate is in PACU until discharged.
Time Frame: Participants will be followed immediately following surgery, approximately 30 minutes. Measurements will be observed immediately following subject's awakening from anesthesia.
Measure: Mean (Standard Deviation); unit: minutes
Arm/Group | Dexmedetomidine | Placebo
Number analyzed (Participants) | 65 | 64
minutes | 21 (9) | 17 (7)

3. Secondary Outcome: Respiratory Complications Peri-Operative
Description: Postoperative adverse respiratory events: moderate to severe coughing, oxygen desaturation (SPO2 <90%), breath holding, bronchospasm, aspiration, stridor and/or laryngospasm during PACU duration to discharge. The adverse respiratory events and the adverse hemodynamic events will be documented by the anesthesia provider in the operating room and by the recovery room nurses in the PACU recovery room. All will be blinded to the drug administered. Measurement will be obtained by "yes"/"no" to each possible adverse respiratory event by anesthesia staff.
Time Frame: Participants will be followed for the duration immediately following surgery, approximately 30 minutes. Measurements will be observed immediately following subject's awakening from anesthesia by Anesthesia staff.
Measure: Mean (Standard Error); unit: events
Arm/Group | Dexmedetomidine | Placebo
Number analyzed (Participants) | 65 | 64
events | 0 (0) | 0 (0)

4. Secondary Outcome: Hemodynamic Instability
Description: Postoperative adverse hemodynamic events: bradycardia-a decrease in heart rate, hypotension-a decrease in systolic blood pressure (both determined as a 30% decrease from baseline) during PACU duration to discharge. The adverse hemodynamic events will be documented by the anesthesia provider in the operating room and by the recovery room nurses in the PACU recovery room. All will be blinded to the drug administered.Measurement will be obtained by "yes"/"no" to each possible adverse respiratory event by anesthesia staff.
Time Frame: as for outcome 3
Measure: Mean (Standard Deviation); unit: events
Arm/Group | Dexmedetomidine | Placebo
Number analyzed (Participants) | 65 | 64
events | 0 (0) | 0 (0)

5. Secondary Outcome: Post-Operative Behavioral Disturbances
Description: Behavioral disturbances analyzed are: sleep disturbances, anxiety, eating disturbances. These post-operative behavioral disturbances are not considered an adverse event. Data regarding postoperative behavioral disturbances will be collected by a blinded individual in a telephone interview 3 days after the surgery. Any "other adverse event" (not including serious) will also be documented by the telephone interview. Measurement will be obtained by "yes"/"no" to each possible AE by staff based on parent(s) response. "Other adverse events" (not including serious) reported immediately post-operatively includes: 1. allergic reaction to medication, 2. Respiratory distress, 3. Bronchospasms 4. Laryngospasm, 5. Hemodynamic instability
Time Frame: Participants will be followed for the duration immediately following surgery, approximately 30 minutes, through approximately Day 3 post-surgery. Measurements will be observed immediately following subject's awakening from anesthesia by Anesthesia staff.
Measure: Number; unit: events
Arm/Group | Dexmedetomidine | Placebo
Number analyzed (Participants) | 65 | 64
events | 9 | 10

6. Secondary Outcome: Muscle Pain
Description: Postoperative muscle pain or swelling at the drug injection site. The duration of the stay in the PACU will be retrospectively documented by the research team using EPIC. Data regarding postoperative muscle pain or swelling will be collected by a blinded individual in a telephone interview 3 days after the surgery. Any adverse event will also be documented by the telephone interview. Measurement will be obtained by "yes"/"no" by staff based on parent(s) response.
Time Frame: as for outcome 5
Measure: Number; unit: events
Arm/Group | Dexmedetomidine | Placebo
Number analyzed (Participants) | 65 | 64
events | 0 | 0

ADVERSE EVENTS:
Time Frame: Participants will be followed for the duration to include immediately following surgery (approximately 30 minutes) through approximately Day 3 post surgery. Measurements will be observed immediately following subject's awakening from anesthesia by anesthesia staff.
Description: Other adverse events (not including serious) reported immediately post-operatively includes: 1. allergic reaction to medication, 2. Respiratory distress, 3. Bronchospasms 4. Laryngospasm, 5. Hemodynamic instability
Arm/Group | Dexmedetomidine | Placebo
All-Cause Mortality (participants affected / at risk) | 0/65 | 0/64
Serious Adverse Events (participants affected / at risk) | 0/65 | 0/64
Other Adverse Events (participants affected / at risk) | 0/65 | 0/64

LIMITATIONS AND CAVEATS:
There were no limitations or caveats that prevented us from completion of the study.

CERTAIN AGREEMENTS:
Principal investigators are sponsor employees: No; Agreement restricts PI disclosure of results: No